CLINICAL TRIAL: NCT05318248
Title: The Role of Stress Neuromodulators in Decision Making Under Risk
Brief Title: The Role of Stress Neuromodulators in Decision Making Under Risk (Part II)
Acronym: SID2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Katja Wingenfeld, Prof. Dr., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: WI 3396-11
Record Dates: First submitted 2022-03-16; First posted 2022-04-08 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Stress
MeSH Terms: interventions — Clonidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clonidin (Experimental): pill 0,15 mg clonidin
  Interventions: Drug: Clonidin
- Placebo (Placebo Comparator): placebo pill
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clonidin — 0,15mg Clonidin orally versus placebo pill
  Arms: Clonidin
Drug: Placebo — placebo pill
  Arms: Placebo

SUMMARY:
The aim of the proposed project is to combine precise pharmacological manipulation of the noradrenergic system with behavioral modeling of memory processes, and fMRI methods to study the effect of a pharmacologically induced blockade of the noradrenergic system on memory processes. Behaviorally, the investigators will focus on the effect of the noradrenergic blockade on working memory performance, and recognition memory.

DETAILED DESCRIPTION:
Affective states like acute stress can influence cognition, i.e., memory processes. Physiologically, acute stress elicits an array of autonomic and endocrine responses, including a fast release of norepinephrine from the locus coeruleus noradrenergic (LC NA) system. Compelling evidence shows that in healthy humans, stimulation of the noradrenergic system increases memory performance whereas noradrenergic blockade reduces memory performance. Functional magnetic resonance imaging (fMRI) studies have shown that manipulations of the noradrenergic system affects responsiveness and connectivity within networks that are important for autonomic-neuroendocrine control and temporal and spatial attention orientation. So far, no study investigated the neural underpinnings of memory processes after a pharmacologically induced noradrenergic blockade. The aim of the proposed project is to combine precise pharmacological manipulation of the noradrenergic system with behavioral modeling of distinct memory processes, and fMRI methods to study the effect of a pharmacologically induced blockade of the noradrenergic system on two distinct memory processes. Behaviorally, the investigators will focus on the effect of the noradrenergic blockade on working memory performance, and recognition memory. Participants are randomly assigned to one of two groups: (A) clonidine, or (B) placebo.

ELIGIBILITY:
Inclusion Criteria:

* right handed, high-school diploma

Exclusion Criteria:

* former & present DSM-5 axis I disorders, medication,

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 82 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Working Memory (n-back task) | 11 minutes
  Behavioral outcome of emotional two-back task = number of correct answers / button presses
Recognition Memory (word list learning) | 25 minutes
  Behavioral outcome of word recognition task = number of correctly recognized words
Blood-oxygen-level-dependent (BOLD) response | 46 minutes
  fMRI data

SECONDARY OUTCOMES:
blood pressure | 2.5 hours
  Treatment check
Heart rate | 2.5 hours
  Treatment check
salivary cortisol | 2.5 hours
  Treatment check

CONTACTS AND LOCATIONS:
Locations (1):
- Charite University, Berlin, Germany